CLINICAL TRIAL: NCT07239622
Title: Liposomal Irinotecan Combined With Sintilimab and Anlotinib in the Treatment of Recurrent or Persistent Ovarian Clear Cell Carcinoma: A Multicenter, Single-Arm, Phase II Clinical Study
Brief Title: Liposomal Irinotecan Combined With Sintilimab and Anlotinib in the Treatment of Recurrent or Persistent Ovarian Clear Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Lu Huaiwu, Department of Gynecological Oncology, Sun Yat-sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, China., Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2025-677-01
Record Dates: First submitted 2025-11-13; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Ovarian Cancer; Ovarian Clear Cell Carcinoma
Keywords: ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): **Treatment Regimen:**
  Participants will receive the following treatment:
  * **Liposomal irinotecan:** Initial dose of 50 mg/m²; if well tolerated, the dose will be increased to 70 mg/m² in subsequent cycles. Administered via intravenous infusion on Day 1 of each 3-week cycle.
  * **Sintilimab:** 200 mg administered by intravenous infusion (over 30-60 minutes) on Day 1 of each cycle.
  * **Anlotinib:** 8 mg orally once daily, starting on Day 1 of each cycle, taken for 2 consecutive weeks followed by a 1-week rest period.
  Interventions: Drug: Treatment

INTERVENTIONS:
Drug: Treatment — Participants will receive the following treatment:
  Liposomal irinotecan: Initial dose of 50 mg/m²; if well tolerated, the dose will be increased to 70 mg/m² in subsequent cycles. Administered via intravenous infusion on Day 1 of each 3-week cycle.
  Sintilimab: 200 mg administered by intravenous infusion (over 30-60 minutes) on Day 1 of each cycle.
  Anlotinib: 8 mg orally once daily, starting on Day 1 of each cycle, taken for 2 consecutive weeks followed by a 1-week rest period.

SUMMARY:
**Primary Objective:** The primary objective of this study is to evaluate the efficacy and safety of liposomal irinotecan in combination with sintilimab and anlotinib in patients with recurrent or persistent ovarian clear cell carcinoma (OCCC).

**Treatment Regimen:**

Participants will receive the following treatment:

* **Liposomal irinotecan:** Initial dose of 50 mg/m²; if well tolerated, the dose will be increased to 70 mg/m² in subsequent cycles. Administered via intravenous infusion on Day 1 of each 3-week cycle.
* **Sintilimab:** 200 mg administered by intravenous infusion (over 30-60 minutes) on Day 1 of each cycle.
* **Anlotinib:** 8 mg orally once daily, starting on Day 1 of each cycle, taken for 2 consecutive weeks followed by a 1-week rest period.

**Follow-up Schedule:** Patients will be followed every 3 months during treatment and within the first year after completion of therapy, every 6 months from Year 2 to Year 5, and annually thereafter. Follow-up assessments will include physical examination, laboratory testing, and imaging studies.

DETAILED DESCRIPTION:
**(1)** This study plans to enroll **36 patients** with recurrent or persistent ovarian clear cell carcinoma (OCCC). Patients who meet all inclusion criteria and do not meet any exclusion criteria will be enrolled in the study.

**(2) Treatment regimen: liposomal irinotecan + sintilimab + anlotinib**

* **Liposomal irinotecan:** Initial dose 50 mg/m²; if well tolerated, increased to 70 mg/m² at the next cycle.

Administered once every 3 weeks (Q3W), intravenous infusion on Day 1 of each cycle.

* **Sintilimab:** 200 mg, intravenous infusion (30-60 minutes), Day 1 of each cycle.
* **Anlotinib:** 8 mg orally, starting on Day 1 of each cycle, administered for 2 weeks followed by 1 week off.

**Administration sequence:** On Day 1 of each cycle, medications are administered in sequence: patients take anlotinib capsules orally while fasting, followed by intravenous infusion of sintilimab. After an interval of at least 30 minutes, liposomal irinotecan is administered intravenously.

Patients will continue treatment until disease progression, unacceptable toxicity, initiation of new anticancer therapy, withdrawal of informed consent, loss to follow-up, death, or other conditions requiring treatment discontinuation per protocol.

If anlotinib must be temporarily or permanently discontinued due to intolerable toxicity during combination therapy, patients may continue sintilimab and liposomal irinotecan until disease progression, unacceptable toxicity, initiation of new therapy, withdrawal of consent, loss to follow-up, death, or termination by the investigator or sponsor.

If sintilimab must be temporarily or permanently discontinued due to intolerable toxicity, patients may continue anlotinib and liposomal irinotecan under the same termination conditions.

If liposomal irinotecan must be temporarily or permanently discontinued due to intolerable toxicity, patients may continue anlotinib and sintilimab under the same termination conditions.

This study aims to evaluate the **efficacy and safety** of sintilimab combined with anlotinib and liposomal irinotecan in patients with histologically confirmed platinum-resistant recurrent or persistent OCCC.

After completing all patient evaluations, a trained study coordinator will introduce the study protocol to potentially eligible participants and provide counseling. Patients who voluntarily agree to participate will be informed of all study details, after which written informed consent will be obtained. Baseline characteristics will be collected from all consented patients, who will then receive sintilimab, anlotinib, and liposomal irinotecan therapy. Subsequent treatment will follow standard clinical practice.

After completion of treatment, patients will be followed every **3 months during the first year**, **every 6 months during years 2-5**, and **annually thereafter**. Follow-up assessments will be conducted during each scheduled visit.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily agrees to participate in the clinical study and signs a written informed consent form.
* Age between 18 and 75 years, with histologically confirmed recurrent or persistent ovarian clear cell carcinoma.
* Has received at least one prior line of platinum-based chemotherapy.
* ECOG performance status of 0-2.
* Expected survival greater than 12 weeks.
* Has measurable disease as defined by RECIST version 1.1:
* Each lesion must measure ≥10 mm in its longest diameter by CT, MRI, or clinical examination;
* Lesions measured by chest X-ray must be ≥20 mm;
* Lymph nodes must have a short axis ≥15 mm when measured by CT or MRI.
* At least 4 weeks have elapsed since the last systemic anticancer therapy.
* Hematologic, hepatic, renal, thyroid, and cardiac enzyme tests are within normal limits.

Exclusion Criteria:

* Non-clear cell histologic subtype of ovarian carcinoma.
* Prior treatment with immune checkpoint inhibitors, including PD-1, PD-L1, or CTLA-4 inhibitors.
* Contraindications to anlotinib, including but not limited to: history of gastrointestinal perforation; surgery within 28 days before combination therapy or unhealed wounds; severe bleeding or recent hemoptysis; or any other condition deemed unsuitable for anlotinib use by the investigator.
* Known allergy to irinotecan, anlotinib, or sintilimab.
* Brain metastases requiring surgical intervention.
* History of other malignancies within the past 5 years.
* Active autoimmune disease within the past 2 years.
* Vaccination within 1 month prior to study enrollment.
* Blood transfusion or platelet transfusion within 4 weeks before first dosing.
* Systemic corticosteroid therapy (excluding topical, inhaled, or intranasal corticosteroids) or any other form of immunosuppressive therapy (e.g., cyclophosphamide, azathioprine, methotrexate, thalidomide, or anti-TNF agents) within 7 days prior to first dosing.
* Use of systemic antitumor traditional Chinese medicine or immunomodulatory agents (e.g., thymosin, interferon, interleukin) within 2 weeks before first dosing, except for local use to control pleural effusion.
* Continuous use of aspirin (>325 mg/day) or other nonsteroidal anti-inflammatory drugs known to inhibit platelet function for 10 consecutive days within 10 days before first dosing.
* Continuous full-dose oral or parenteral anticoagulant or thrombolytic therapy for 10 consecutive days within 10 days before first dosing.
* Hereditary bleeding tendency or coagulation disorder; history of hypertension with thrombosis; tumor invasion of major vessels, or radiologic evidence suggesting risk of bleeding, as determined by the investigator or radiologist.
* Presence of serious unhealed wounds, ulcers, or fractures.
* History of allogeneic organ transplantation (except corneal transplant) or allogeneic hematopoietic stem cell transplantation.
* Known history of human immunodeficiency virus (HIV) infection (positive HIV-1/2 antibodies).
* Untreated active hepatitis B infection (defined as HBsAg positive with detectable HBV-DNA copies).
* Unresolved toxicities from prior therapy (≥Grade 2), except for alopecia, neuropathy, lymphopenia, or skin depigmentation.
* Presence of severe or uncontrolled systemic diseases

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Patients will be followed every 3 months during treatment and up to 1 year after treatment completion, every 6 months from Year 2 to Year 5, and annually thereafter (up to 6 years).
  ORR is defined as the proportion of patients whose tumors have shrunk to a predefined extent, including cases achieving complete response (CR) or partial response (PR). Tumor response will be assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
  Measurable lesions will be documented before treatment initiation, and tumor assessments will be performed every two treatment cycles to evaluate changes until disease progression or treatment discontinuation.
  According to RECIST v1.1, treatment response will be categorized as:
  Complete Response (CR): Disappearance of all target lesions.
  Partial Response (PR): ≥30% decrease in the sum of diameters of target lesions.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
  Progressive Disease (PD): ≥20% increase in the sum of diameters of target lesions or the appearance of new lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Huaiwu Lu, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University

IPD SHARING:
Plan to Share IPD: No